CLINICAL TRIAL: NCT07134530
Title: Advanced Cardiovascular Management in Major Non-cardiac Surgery. A Single Center, Randomized, Parallel, Open Label Clinical Trial
Brief Title: Advanced Cardiovascular Management in Major Non-cardiac Surgery.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Alessandro Locatelli, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIMS
Record Dates: First submitted 2025-08-12; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Intraoperative Hypotension
Keywords: Intraoperative hypotension; major non-cardiac surgery; IOH; Acumen Hypotension Prediction Index (HPI) system

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-risk adult patients undergoing major non cardiac surgery (Active Comparator): Standard GDT strategy
  Interventions: Device: GDT strategy
- high-risk adult patients undergoing major non cardiac surgery (Experimental): HPI-driven intraoperative hemodynamic management strategy
  Interventions: Device: HPI-driven intraoperative hemodynamic management strategy

INTERVENTIONS:
Device: HPI-driven intraoperative hemodynamic management strategy — Hemodynamic management protocol based on information detected by Edwards HemoSphere monitor equipped with the Acumen Hypotension Prediction Index software (HPI)
Device: GDT strategy — Current clinical hemodynamic care

SUMMARY:
This is a single center, randomised and controlled clinical triaI whose aim is to predict and treat in advance, intraoperative hypotension episodes.

In particular, the aim of the study is to compare the clinical impact of two different hemodynamic strategies based on the use of different monitoring platforms: the Edwards EV1000 equipped with FloTrac sensor and HemoSphere platform equipped with Acumen Hypotension Prediction Index software and Acumen IQ pressure sensor.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Age ≥ 18 years old
* Surgical indication for major NCS needing general anesthesia
* Anaesthesiologic indication for perioperative arterial cannulation and advanced hemodynamic monitoring

Exclusion Criteria:

* Informed Refusal as documented by signature (Appendix Informed Consent Form)
* Age ≤ 18 years old
* Severe aortic valvulopathy
* Atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
MINS and AKI incidence | within 3 and 7 days after surgery
  Clinical impact of any reduction in IOH occurrence or severity

SECONDARY OUTCOMES:
Mortality | 30 days
Cardiac damage | from day 1 to 3
  Measure of serum high-specific Troponin I
kidney damage | day 1, day 2 and day 7
  measure of creatine
hypotensive events | 2 years
  severity and time-weighted average

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Pavia, Italy